CLINICAL TRIAL: NCT06336148
Title: A Phase 1a/1b Open-label, Dose-Escalation and Expansion Study of ACTM-838 as a Single Agent in Patients With Advanced Solid Tumors
Brief Title: A Phase 1a/1b Study of ACTM-838 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's strategic business decision
Sponsor: Actym Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTM-838-01
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor
Keywords: non-small cell lung cancer; head and neck cancer; esophageal cancer; ovarian cancer; cervical cancer; stomach cancer; thyroid cancer; renal cell cancer; mesothelioma; breast cancer; pancreatic cancer; colorectal cancer; sarcoma; immunotherapy; melanoma; bladder cancer; cholangiocarcinoma; bile duct cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms; Esophageal Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Stomach Neoplasms; Thyroid Neoplasms; Carcinoma, Renal Cell; Mesothelioma; Breast Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Sarcoma; Melanoma; Urinary Bladder Neoplasms; Cholangiocarcinoma; Bile Duct Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an Open label Single dose study.
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACTM-838 Monotherapy (Experimental): Escalating doses of ACTM-838 in Part 1a followed by expansion in Part 1b at the recommended dose determined in Part 1a
  Interventions: Drug: ACTM-838

INTERVENTIONS:
Drug: ACTM-838 — Escalating doses of ACTM-838 in Part 1a and recommended dose in Part 1b

SUMMARY:
This is a first in human (FIH) 2-part study using ACTM-838 in patients with advanced solid tumors resistant to standard of care treatment. Part 1a will evaluate dose escalation and Part 1b will evaluate dose expansion.

DETAILED DESCRIPTION:
This study has 2 parts. Part 1a will evaluate the safety and tolerability and activity of escalating doses of ACTM-838 to estimate the maximum tolerated dose (MTD) and/or the optimum biological dose (OBD) for ACTM-838 as a monotherapy and determine the dose recommended for Part 1b.

Part 1b will further evaluate ACTM-838 in patients with advanced specific tumor types (defined pathologically, clinically and/or molecularly) based on data emerging from the Phase 1a and the pre-clinical program. The details on the Phase 1b dose expansion part will be incorporated in a future protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced solid tumor for which there is no remaining standard curative therapy and no therapy with a demonstrated survival benefit, or they must be ineligible to receive or refuse to receive such therapy
2. At least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST ) v1.1; amenable for biopsy, and radiographically apparent on computed tomography (CT) or magnetic resonance imaging (MRI )
3. Eastern Cooperative Oncology Group (ECOG) 0-1
4. Adequate hematologic, hepatic, pulmonary, and cardiac function
5. CD4 count >500/mL at screening
6. Additional protocol defined inclusion criteria may apply

Exclusion Criteria:

1. Active autoimmune disease requiring systemic treatment (i.e., with use of disease modifying agents, systemic corticosteroids or immunosuppressive drug) within the past 6 months prior to dosing of investigational product.
2. History of permanent artificial implants (e.g., prosthetic joints, artificial heart valves, pacemakers, orthopaedic screw[s], metal plate[s], bone graft[s], or other exogenous implant[s]
3. Known history of cholelithiasis or urolithiasis
4. History of valvular disease, arterial aneurisms or arterial or venous malformation
5. Known active brain metastases
6. Documented active Salmonella infection or vaccination with Salmonella typhi within 6 months prior to investigational product dosing
7. Additional protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and serious adverse events - Part 1a | 1 year
Proportion of participants experiencing dose limiting toxicities - Part 1a | 28 Days

SECONDARY OUTCOMES:
Objective response rate (ORR) defined as complete response (CR) or partial response (PR) - Part 1a | 1 year
Confirmed ORR defined as confirmed CR or confirmed PR - Part 1a | 1 year
Clinical Benefit Rate (CR, PR, or stable disease (SD) as best overall response) - Part 1a | 1 year
Duration of Response (DoR), defined as the time from date of first response (CR or PR) - Part 1a | 1 year
Progression free survival (PFS) - Part 1a | 1 year
Change in tumor markers - Part 1a | 1 year
Amount of ACTM-838 in blood, urine, and faeces as measured by digital droplet-polymerase chain reaction (ddPCR) - Part 1a | 1 year
Tumor PD colonization as measured by ddPCR and payload delivery as measured by RNA detection - Part 1a | 1 year
Incidence of antidrug antibodies (ADA) to ACTM-838 - Part 1a | 1 year

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - University of Southern California Norris Comprehensive Cancer Center, 1441 Eastlake Ave., Los Angeles, California
  - UPMC Hillman Cancer Center, 5115 Centre Ave, Pittsburgh, Pennsylvania
- Australia (3):
  - Westmead Hospital, Cnr Hawkesbury Road and Darcy Road, Site No: 200, Westmead, New South Wales
  - Southern Oncology Clinical Research Unit, Level 3, Mark Oliphant Building, 5 Laffer Drive, Site No: 202, Bedford Park, South Australia
  - Alfred Hospital, 55 Commercial Road, Site No: 201, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No